CLINICAL TRIAL: NCT05804669
Title: A Phase 1b/2a Open-label Multiple-ascending Dose Exploratory Study of CRN04894 in ACTH-dependent Cushing's Syndrome (Cushing's Disease or Ectopic ACTH Syndrome)
Brief Title: A Study to Evaluate the Safety and PK of CRN04894 for the Treatment of Cushing's Syndrome
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRN04894-04
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Cushing Syndrome; Cushing Disease; Ectopic ACTH Syndrome
Keywords: Cushing Syndrome; Cushing Disease; Ectopic ACTH Syndrome; CRN04894; atumelnant
MeSH Terms: conditions — Cushing Syndrome; Pituitary ACTH Hypersecretion; ACTH Syndrome, Ectopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multiple Ascending Doses (Experimental): Sequential, open-label, 10-day or 14-day fixed-dose cohorts.
  Interventions: Drug: atumelnant

INTERVENTIONS:
Drug: atumelnant — Atumelnant is an orally active investigational agent which antagonizes the action of ACTH at its receptor administered as oral tablets.

SUMMARY:
A Phase 1b/2a, first-in-disease, open-label, multiple-ascending dose exploratory study to evaluate safety, tolerability, pharmacokinetics (PK), and pharmacodynamic biomarker responses associated with CRN04894 (an adrenocorticotropic hormone [ACTH] receptor antagonist) in participants with ACTH-dependent Cushing's syndrome (Cushing's disease or Ectopic ACTH Syndrome [EAS])

DETAILED DESCRIPTION:
This is a Phase 1b/2a, first-in-disease, open-label, multiple-ascending dose exploratory study to evaluate safety, tolerability, pharmacokinetics (PK), and pharmacodynamic biomarker responses associated with atumelnant (also known as CRN04894) (an adrenocorticotropic hormone [ACTH] receptor antagonist) over a 10-day or 14-day treatment period in participants with ACTH-dependent Cushing's syndrome (Cushing's disease or Ectopic ACTH Syndrome [EAS]). Participants will receive oral atumelnant once daily for 10 days followed by monitoring during 4 'wash-out' days, or for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female, aged 18 years or more
2. Evidence of chronic 'active' ACTH-dependent Cushing's syndrome
3. Evidence of acutely 'active' ACTH-dependent Cushing's syndrome within 10 days of Day 1
4. Participants with documented ACTH-dependent Cushing's syndrome taking short-acting steroidogenesis inhibitors (ketoconazole, levoketoconazole, osilodrostat, or metyrapone) may participate after a washout period of at least 5 days, if they meet other study inclusion criteria, relative to Investigator's judgment. Participants with documented ACTH-dependent Cushing's syndrome taking cabergoline may participate after a washout period of at least 14 days, if they meet other study inclusion criteria

Exclusion Criteria:

1. Women who are pregnant or lactating
2. History of bilateral adrenalectomy
3. Previous pituitary MRI findings of a putative ACTH-secreting lesion within 3 mm of the optic chiasm
4. Presence of any known malignancy
5. Use of mitotane
6. Previous unsuccessful surgery for Cushing's syndrome within 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with treatment emergent adverse events (TEAEs) | Up to Day 15
Proportion of participants with adrenal insufficiency | Up to Day 15
Proportion of participants with safety findings determined by laboratory testing | Up to Day 15
Assessment of the maximum observed plasma concentration of CRN04894 | Up to Day 15
Assessment of the time to achieve maximum observed plasma concentration of CRN04894 | Up to Day 15
Assessment of the plasma area under the curve of CRN04894 | Up to Day 15

SECONDARY OUTCOMES:
Change from baseline in early morning serum cortisol | Up to Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health (NIH) - National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No